CLINICAL TRIAL: NCT02074631
Title: Prevention of Bone Loss After Pediatric Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013LS023
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Osteopenia; Osteoporosis
Keywords: bone mineral content; bone mineral density; bone formation; bone resorption; pamidronate; children; DXA; bone marrow transplant
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Bone Resorption | interventions — Pamidronate; Calcium; Vitamin D; Cholecalciferol; Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Subjects will receive a standard recommended dose of calcium and vitamin D.
  Interventions: Drug: Calcium and vitamin D
- Pamidronate Group (Experimental): Subjects randomized to pamidronate treatment will receive infusions approximately 100, 180, and 270 days after HCT along with calcium and vitamin D.
  Interventions: Drug: Pamidronate; Drug: Calcium and vitamin D

INTERVENTIONS:
Drug: Pamidronate — Subjects randomized to pamidronate treatment will receive infusions, 1 mg/kg (to a max dose of 60mg) over 4 hours, every 3 months at approximately 100 days, 180 days, and 270 days after HCT.
  Other Names: Aredia; Bonapam
  Arms: Pamidronate Group
Drug: Calcium and vitamin D — All subjects will receive a standard recommended dose of 600 IU/day of vitamin D. Subjects who do not meet the RDA will receive additional calcium supplementation.
  Other Names: Cholecalciferol; Ergocalciferol

SUMMARY:
This is a Phase 2, open-label, randomized, controlled clinical study of pediatric subjects treated with pamidronate with calcium and vitamin D versus calcium and vitamin D alone following hematopoietic cell transplantation (HCT). The purpose of this study is to test the hypothesis that subjects receiving pamidronate with calcium and vitamin D will have higher lumbar spine bone mineral content (LBMC) measured by dual-energy X-ray tomography (DXA) at 1 year post-HCT than subjects receiving calcium and vitamin D alone (Control Group).

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic hematopoietic cell transplant for hematologic malignancy (i.e. leukemia, lymphoma including ALL, AML, CML, NHL, HL) in complete remission; myelodysplastic syndrome (active dysplasia and/or blasts are permitted, but must not have active leukemia) or idiopathic severe aplastic anemia (SAA)
* Non-malignant diseases including idiopathic severe aplastic anemia (SAA) and other bone marrow failure disorders, hemoglobinopathies, adrenoleukodystrophy, immune deficiencies/dysregulation disorders who will be receiving myeloablative or reduced toxicity preparative regimens that meet the following criteria:

  * Regimens include those that are TBI based if the TBI dose is > 500cGy single dose or > 800cGy fractionated, or doses <500 cGy if combined with busulfan or treosulfan. These also include chemotherapy only based regimens that contain myeloablative doses of busulfan (>8mg/kg) or treosulfan without TBI.
  * Patients with severe aplastic anemia are eligible regardless of conditioning regimen
* Myeloablative preparative regimen (for SAA any conditioning therapy allowed)
* Male or female ≥1 but ≤ 20 years of age at time of study enrollment
* Patient or parent(s)/legal guardian(s) is able and willing to provide informed consent. Assent will be obtained per local institutional policy. Subjects who turn 18 during the course of the study will be consented at that time of their next visit by a member of the research staff.

Exclusion Criteria:

* History of a primary bone malignancy involving the lumbar spine
* Prior and/or planned concomitant medical therapy during the study period (through Day 360 post-HCT) with other bisphosphonates, Denosumab, or Teriparatide
* Pregnancy or breastfeeding - menstruating females must have a negative pregnancy test prior to study enrollment and agree to repeat pregnancy testing and contraception use per protocol as pamidronate is Pregnancy Category D - positive evidence of human fetal risk based on adverse reaction data
* Renal insufficiency, defined as creatinine level greater than the upper limit of normal for age
* Hereditary metabolic bone disease or skeletal dysplasia (e.g., osteopetrosis or OI) or primary hyperparathyroidism
* Other indications for HCT, including Fanconi anemia, other form of inherited bone marrow failure diseases, metabolic disorder, hemoglobinopathy, or immune deficiency
* Clinically significant fractures as defined by ISCD (a long bone fracture of the lower extremities, vertebral compression fracture, or two or more long bone fractures of the upper extremities) (88,89) indicated by a cast or a spine x-ray within the last 2 weeks
* Known or suspected allergy to pamidronate or related products
* Planned administration of an investigational study drug or agent that either can interact with pamidronate or have an independent effect on bone mineral density within the 4 weeks prior to randomization (Day 90) or planned use during study participation (Day 90 through Day 360)
* Impending invasive dental procedure that would be expected to occur during study participation (through Day 360)

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakie Sarafoglou, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Amplatz Children's Hospital, Minneapolis, Minnesota
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Petryk A, Bergemann TL, Polga KM, Ulrich KJ, Raatz SK, Brown DM, Robison LL, Baker KS. Prospective study of changes in bone mineral density and turnover in children after hematopoietic cell transplantation. J Clin Endocrinol Metab. 2006 Mar;91(3):899-905. doi: 10.1210/jc.2005-1927. Epub 2005 Dec 13. PMID 16352681
- [Background] Bhatia S, Ramsay NK, Weisdorf D, Griffiths H, Robison LL. Bone mineral density in patients undergoing bone marrow transplantation for myeloid malignancies. Bone Marrow Transplant. 1998 Jul;22(1):87-90. doi: 10.1038/sj.bmt.1701275. PMID 9678801
- [Background] Nysom K, Holm K, Michaelsen KF, Hertz H, Jacobsen N, Muller J, Molgaard C. Bone mass after allogeneic BMT for childhood leukaemia or lymphoma. Bone Marrow Transplant. 2000 Jan;25(2):191-6. doi: 10.1038/sj.bmt.1702131. PMID 10673679
- [Background] Kaste SC, Shidler TJ, Tong X, Srivastava DK, Rochester R, Hudson MM, Shearer PD, Hale GA. Bone mineral density and osteonecrosis in survivors of childhood allogeneic bone marrow transplantation. Bone Marrow Transplant. 2004 Feb;33(4):435-41. doi: 10.1038/sj.bmt.1704360. PMID 14716354
- [Background] Perkins JL, Kunin-Batson AS, Youngren NM, Ness KK, Ulrich KJ, Hansen MJ, Petryk A, Steinberger J, Anderson FS, Baker KS. Long-term follow-up of children who underwent hematopoeitic cell transplant (HCT) for AML or ALL at less than 3 years of age. Pediatr Blood Cancer. 2007 Dec;49(7):958-63. doi: 10.1002/pbc.21207. PMID 17474113
- [Background] Daniels MW, Wilson DM, Paguntalan HG, Hoffman AR, Bachrach LK. Bone mineral density in pediatric transplant recipients. Transplantation. 2003 Aug 27;76(4):673-8. doi: 10.1097/01.TP.0000076627.70050.53. PMID 12973107
- [Background] Mostoufi-Moab S, Ginsberg JP, Bunin N, Zemel B, Shults J, Leonard MB. Bone density and structure in long-term survivors of pediatric allogeneic hematopoietic stem cell transplantation. J Bone Miner Res. 2012 Apr;27(4):760-9. doi: 10.1002/jbmr.1499. PMID 22189761
- [Background] Jackowski SA, Kontulainen SA, Cooper DM, Lanovaz JL, Baxter-Jones AD. The timing of BMD and geometric adaptation at the proximal femur from childhood to early adulthood in males and females: a longitudinal study. J Bone Miner Res. 2011 Nov;26(11):2753-61. doi: 10.1002/jbmr.468. PMID 21773991
- [Background] Kaste SC, Rai SN, Fleming K, McCammon EA, Tylavsky FA, Danish RK, Rose SR, Sitter CD, Pui CH, Hudson MM. Changes in bone mineral density in survivors of childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2006 Jan;46(1):77-87. doi: 10.1002/pbc.20553. PMID 16106430
- [Background] Ross PD, Davis JW, Epstein RS, Wasnich RD. Pre-existing fractures and bone mass predict vertebral fracture incidence in women. Ann Intern Med. 1991 Jun 1;114(11):919-23. doi: 10.7326/0003-4819-114-11-919. PMID 2024857
- [Background] Baxter-Jones AD, Faulkner RA, Forwood MR, Mirwald RL, Bailey DA. Bone mineral accrual from 8 to 30 years of age: an estimation of peak bone mass. J Bone Miner Res. 2011 Aug;26(8):1729-39. doi: 10.1002/jbmr.412. PMID 21520276
- [Background] Polgreen LE, Rudser K, Deyo M, Smith A, Baker KS, Petryk A. Changes in biomarkers of bone resorption over the first six months after pediatric hematopoietic cell transplantation. Pediatr Transplant. 2012 Dec;16(8):852-7. doi: 10.1111/j.1399-3046.2012.01780.x. Epub 2012 Aug 20. PMID 22905997
- [Background] Grigg AP, Shuttleworth P, Reynolds J, Schwarer AP, Szer J, Bradstock K, Hui C, Herrmann R, Ebeling PR. Pamidronate reduces bone loss after allogeneic stem cell transplantation. J Clin Endocrinol Metab. 2006 Oct;91(10):3835-43. doi: 10.1210/jc.2006-0684. Epub 2006 Jul 11. PMID 16835281
- [Background] Kananen K, Volin L, Laitinen K, Alfthan H, Ruutu T, Valimaki MJ. Prevention of bone loss after allogeneic stem cell transplantation by calcium, vitamin D, and sex hormone replacement with or without pamidronate. J Clin Endocrinol Metab. 2005 Jul;90(7):3877-85. doi: 10.1210/jc.2004-2161. Epub 2005 Mar 29. PMID 15797959
- [Background] Glorieux FH. Treatment of osteogenesis imperfecta: who, why, what? Horm Res. 2007;68 Suppl 5:8-11. doi: 10.1159/000110463. Epub 2007 Dec 10. PMID 18174695
- [Background] Land C, Rauch F, Travers R, Glorieux FH. Osteogenesis imperfecta type VI in childhood and adolescence: effects of cyclical intravenous pamidronate treatment. Bone. 2007 Mar;40(3):638-44. doi: 10.1016/j.bone.2006.10.010. Epub 2006 Nov 28. PMID 17127117
- [Background] Devogelaer JP, Malghem J, Maldague B, Nagant de Deuxchaisnes C. Radiological manifestations of bisphosphonate treatment with APD in a child suffering from osteogenesis imperfecta. Skeletal Radiol. 1987;16(5):360-3. doi: 10.1007/BF00350961. PMID 3629280
- [Background] Rauch F, Glorieux FH. Osteogenesis imperfecta. Lancet. 2004 Apr 24;363(9418):1377-85. doi: 10.1016/S0140-6736(04)16051-0. PMID 15110498
- [Background] Speiser PW, Clarson CL, Eugster EA, Kemp SF, Radovick S, Rogol AD, Wilson TA; LWPES Pharmacy and Therapeutic Committee. Bisphosphonate treatment of pediatric bone disease. Pediatr Endocrinol Rev. 2005 Dec;3(2):87-96. PMID 16361982
- [Background] Castillo H, Samson-Fang L; American Academy for Cerebral Palsy and Developmental Medicine Treatment Outcomes Committee Review Panel. Effects of bisphosphonates in children with osteogenesis imperfecta: an AACPDM systematic review. Dev Med Child Neurol. 2009 Jan;51(1):17-29. doi: 10.1111/j.1469-8749.2008.03222.x. PMID 19087101
- [Background] DiMeglio LA, Ford L, McClintock C, Peacock M. Intravenous pamidronate treatment of children under 36 months of age with osteogenesis imperfecta. Bone. 2004 Nov;35(5):1038-45. doi: 10.1016/j.bone.2004.07.003. PMID 15542028
- [Background] Glorieux FH, Bishop NJ, Plotkin H, Chabot G, Lanoue G, Travers R. Cyclic administration of pamidronate in children with severe osteogenesis imperfecta. N Engl J Med. 1998 Oct 1;339(14):947-52. doi: 10.1056/NEJM199810013391402. PMID 9753709
- [Background] Henderson RC, Lark RK, Kecskemethy HH, Miller F, Harcke HT, Bachrach SJ. Bisphosphonates to treat osteopenia in children with quadriplegic cerebral palsy: a randomized, placebo-controlled clinical trial. J Pediatr. 2002 Nov;141(5):644-51. doi: 10.1067/mpd.2002.128207. PMID 12410192
- [Background] Plotkin H, Coughlin S, Kreikemeier R, Heldt K, Bruzoni M, Lerner G. Low doses of pamidronate to treat osteopenia in children with severe cerebral palsy: a pilot study. Dev Med Child Neurol. 2006 Sep;48(9):709-12. doi: 10.1017/S0012162206001526. PMID 16904014
- [Background] Grissom LE, Kecskemethy HH, Bachrach SJ, McKay C, Harcke HT. Bone densitometry in pediatric patients treated with pamidronate. Pediatr Radiol. 2005 May;35(5):511-7. doi: 10.1007/s00247-004-1393-3. Epub 2005 Jan 18. PMID 15655696
- [Background] Gandrud LM, Cheung JC, Daniels MW, Bachrach LK. Low-dose intravenous pamidronate reduces fractures in childhood osteoporosis. J Pediatr Endocrinol Metab. 2003 Jul-Aug;16(6):887-92. doi: 10.1515/jpem.2003.16.6.887. PMID 12948302
- [Background] Brumsen C, Hamdy NA, Papapoulos SE. Long-term effects of bisphosphonates on the growing skeleton. Studies of young patients with severe osteoporosis. Medicine (Baltimore). 1997 Jul;76(4):266-83. doi: 10.1097/00005792-199707000-00005. PMID 9279333
- [Background] Przkora R, Herndon DN, Sherrard DJ, Chinkes DL, Klein GL. Pamidronate preserves bone mass for at least 2 years following acute administration for pediatric burn injury. Bone. 2007 Aug;41(2):297-302. doi: 10.1016/j.bone.2007.04.195. Epub 2007 May 8. PMID 17561466
- [Background] Carpenter PA, Hoffmeister P, Chesnut CH 3rd, Storer B, Charuhas PM, Woolfrey AE, Sanders JE. Bisphosphonate therapy for reduced bone mineral density in children with chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2007 Jun;13(6):683-90. doi: 10.1016/j.bbmt.2007.02.001. Epub 2007 Apr 6. PMID 17531778
- [Background] Whyte MP, Wenkert D, Clements KL, McAlister WH, Mumm S. Bisphosphonate-induced osteopetrosis. N Engl J Med. 2003 Jul 31;349(5):457-63. doi: 10.1056/NEJMoa023110. No abstract available. PMID 12890844
- [Background] Rauch F, Plotkin H, Travers R, Zeitlin L, Glorieux FH. Osteogenesis imperfecta types I, III, and IV: effect of pamidronate therapy on bone and mineral metabolism. J Clin Endocrinol Metab. 2003 Mar;88(3):986-92. doi: 10.1210/jc.2002-021371. PMID 12629073
- [Background] Astrom E, Soderhall S. Beneficial effect of long term intravenous bisphosphonate treatment of osteogenesis imperfecta. Arch Dis Child. 2002 May;86(5):356-64. doi: 10.1136/adc.86.5.356. PMID 11970931
- [Background] Steelman J, Zeitler P. Treatment of symptomatic pediatric osteoporosis with cyclic single-day intravenous pamidronate infusions. J Pediatr. 2003 Apr;142(4):417-23. doi: 10.1067/mpd.2003.137. PMID 12712060
- [Background] Ward LM, Denker AE, Porras A, Shugarts S, Kline W, Travers R, Mao C, Rauch F, Maes A, Larson P, Deutsch P, Glorieux FH. Single-dose pharmacokinetics and tolerability of alendronate 35- and 70-milligram tablets in children and adolescents with osteogenesis imperfecta type I. J Clin Endocrinol Metab. 2005 Jul;90(7):4051-6. doi: 10.1210/jc.2004-2054. Epub 2005 Apr 12. PMID 15827104
- [Background] Zacharin M, Bateman J. Pamidronate treatment of osteogenesis imperfecta--lack of correlation between clinical severity, age at onset of treatment, predicted collagen mutation and treatment response. J Pediatr Endocrinol Metab. 2002 Feb;15(2):163-74. doi: 10.1515/jpem.2002.15.2.163. PMID 11874181
- [Background] Janssen van Doorn K, Neyns B, Van der Niepen P, Verbeelen D. Pamidronate-related nephrotoxicity (tubulointerstitial nephritis) in a patient with osteolytic bone metastases. Nephron. 2001 Dec;89(4):467-8. doi: 10.1159/000046123. No abstract available. PMID 11721169
- [Background] Machado CE, Flombaum CD. Safety of pamidronate in patients with renal failure and hypercalcemia. Clin Nephrol. 1996 Mar;45(3):175-9. PMID 8706358
- [Background] Lin JH. Bisphosphonates: a review of their pharmacokinetic properties. Bone. 1996 Feb;18(2):75-85. doi: 10.1016/8756-3282(95)00445-9. PMID 8833200
- [Background] Papapoulos SE, Cremers SC. Prolonged bisphosphonate release after treatment in children. N Engl J Med. 2007 Mar 8;356(10):1075-6. doi: 10.1056/NEJMc062792. No abstract available. PMID 17347467
- [Background] Ward KA, Adams JE, Freemont TJ, Mughal MZ. Can bisphosphonate treatment be stopped in a growing child with skeletal fragility? Osteoporos Int. 2007 Aug;18(8):1137-40. doi: 10.1007/s00198-007-0330-3. Epub 2007 Feb 6. PMID 17279467
- [Background] Rauch F, Cornibert S, Cheung M, Glorieux FH. Long-bone changes after pamidronate discontinuation in children and adolescents with osteogenesis imperfecta. Bone. 2007 Apr;40(4):821-7. doi: 10.1016/j.bone.2006.11.020. Epub 2007 Jan 12. PMID 17223617
- [Background] Whyte MP, McAlister WH, Novack DV, Clements KL, Schoenecker PL, Wenkert D. Bisphosphonate-induced osteopetrosis: novel bone modeling defects, metaphyseal osteopenia, and osteosclerosis fractures after drug exposure ceases. J Bone Miner Res. 2008 Oct;23(10):1698-707. doi: 10.1359/jbmr.080511. PMID 18505375
- [Background] Janz KF, Letuchy EM, Eichenberger Gilmore JM, Burns TL, Torner JC, Willing MC, Levy SM. Early physical activity provides sustained bone health benefits later in childhood. Med Sci Sports Exerc. 2010 Jun;42(6):1072-8. doi: 10.1249/MSS.0b013e3181c619b2. PMID 19997029
- [Background] Meyer U, Romann M, Zahner L, Schindler C, Puder JJ, Kraenzlin M, Rizzoli R, Kriemler S. Effect of a general school-based physical activity intervention on bone mineral content and density: a cluster-randomized controlled trial. Bone. 2011 Apr 1;48(4):792-7. doi: 10.1016/j.bone.2010.11.018. Epub 2010 Dec 15. PMID 21167330
- [Background] Buison AM, Kawchak DA, Schall JI, Ohene-Frempong K, Stallings VA, Leonard MB, Zemel BS. Bone area and bone mineral content deficits in children with sickle cell disease. Pediatrics. 2005 Oct;116(4):943-9. doi: 10.1542/peds.2004-2582. PMID 16199706
- [Background] Burnham JM, Shults J, Semeao E, Foster B, Zemel BS, Stallings VA, Leonard MB. Whole body BMC in pediatric Crohn disease: independent effects of altered growth, maturation, and body composition. J Bone Miner Res. 2004 Dec;19(12):1961-8. doi: 10.1359/JBMR.040908. Epub 2004 Sep 20. PMID 15537438
- [Background] Horlick M, Wang J, Pierson RN Jr, Thornton JC. Prediction models for evaluation of total-body bone mass with dual-energy X-ray absorptiometry among children and adolescents. Pediatrics. 2004 Sep;114(3):e337-45. doi: 10.1542/peds.2004-0301. PMID 15342895
- [Background] Petryk A, Polgreen LE, Zhang L, Hodges JS, Dengel DR, Hoffmeister PA, Steinberger J, Baker KS. Bone mineral deficits in recipients of hematopoietic cell transplantation: the impact of young age at transplant. Bone Marrow Transplant. 2014 Feb;49(2):258-63. doi: 10.1038/bmt.2013.156. Epub 2013 Oct 14. PMID 24121211
- [Background] Marshall WA, Tanner JM. Variations in pattern of pubertal changes in girls. Arch Dis Child. 1969 Jun;44(235):291-303. doi: 10.1136/adc.44.235.291. No abstract available. PMID 5785179
- [Background] Marshall WA, Tanner JM. Variations in the pattern of pubertal changes in boys. Arch Dis Child. 1970 Feb;45(239):13-23. doi: 10.1136/adc.45.239.13. PMID 5440182
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Background] Misra M, Pacaud D, Petryk A, Collett-Solberg PF, Kappy M; Drug and Therapeutics Committee of the Lawson Wilkins Pediatric Endocrine Society. Vitamin D deficiency in children and its management: review of current knowledge and recommendations. Pediatrics. 2008 Aug;122(2):398-417. doi: 10.1542/peds.2007-1894. PMID 18676559
- [Background] Gordon CM, Williams AL, Feldman HA, May J, Sinclair L, Vasquez A, Cox JE. Treatment of hypovitaminosis D in infants and toddlers. J Clin Endocrinol Metab. 2008 Jul;93(7):2716-21. doi: 10.1210/jc.2007-2790. Epub 2008 Apr 15. PMID 18413426
- [Result] Tauchmanova L, Colao A, Lombardi G, Rotoli B, Selleri C. Bone loss and its management in long-term survivors from allogeneic stem cell transplantation. J Clin Endocrinol Metab. 2007 Dec;92(12):4536-45. doi: 10.1210/jc.2006-2870. Epub 2007 Oct 2. PMID 17911175

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Pamidronate Group
Started | 32 | 31
Completed | 30 | 24
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Pamidronate Group | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 30 | 59
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 20 | 16 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 22 | 24 | 46
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Content
Time Frame: 1 year after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: Average grams
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 29 | 23
Average grams | 41.4 (22.8) | 38.7 (22.2)

2. Secondary Outcome: Total Body Bone Mineral Content (TBMC; Excluding Head; Adjusted for Height, Age, Sex, Tanner Stage, and Race)
Time Frame: 1 year after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Error); unit: Average grams
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 28 | 20
Average grams | 1231 (95) | 1204 (113)

3. Secondary Outcome: Total Bone Mineral Density (BMD), Cortical BMD, Trabecular BMD, and Estimated Bone Strength Measured by pQCT
Description: Measured in g/cm2.
Time Frame: 1 year after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 29 | 21
g/cm2 | 0.829 (0.202) | 0.760 (0.189)

4. Secondary Outcome: Cytokine Levels (Interleukin IL-6, IL-7, and TNF-α)
Description: Measured in pg/ml.
Time Frame: 7 days, 14 days, 21 days, 90 days after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 28 | 27
pg/ml
  IL-6 7 days after HCT | 37.4 (46.6) | 41.4 (49.4)
  IL-6 14 days after HCT: number analyzed (Participants) | 27 | 27
  IL-6 14 days after HCT | 23.6 (19.9) | 35.4 (32.7)
  IL-6 21 days after HCT: number analyzed (Participants) | 27 | 23
  IL-6 21 days after HCT | 22.0 (63.9) | 18.1 (17.5)
  IL-6 90 days after HCT: number analyzed (Participants) | 25 | 27
  IL-6 90 days after HCT | 10.7 (33.9) | 6.8 (5.0)
  IL-7 7 days after HCT | 35.8 (15.6) | 33.4 (19.3)
  IL-7 14 days after HCT: number analyzed (Participants) | 27 | 27
  IL-7 14 days after HCT | 33.7 (14.7) | 35.9 (27.4)
  IL-7 21 days after HCT: number analyzed (Participants) | 27 | 23
  IL-7 21 days after HCT | 28.8 (15.7) | 31.5 (25.9)
  IL-7 90 days after HCT: number analyzed (Participants) | 25 | 27
  IL-7 90 days after HCT | 11.4 (9.5) | 13.1 (11.6)
  TNFa 7 days after HCT | 7.0 (2.8) | 6.9 (3.4)
  TNFa 14 days after HCT: number analyzed (Participants) | 27 | 27
  TNFa 14 days after HCT | 10.5 (5.6) | 11.4 (9.4)
  TNFa 21 days after HCT: number analyzed (Participants) | 27 | 23
  TNFa 21 days after HCT | 11.3 (5.7) | 12.7 (7.2)
  TNFa 90 days after HCT: number analyzed (Participants) | 25 | 27
  TNFa 90 days after HCT | 14.3 (6.5) | 15.9 (7.5)

5. Secondary Outcome: Receptor Activator of the Nuclear Factor-κB Ligand [RANKL], Osteoprotegerin [OPG]
Description: Measured in pg/ml.
Time Frame: 7 days, 14 days, 21 days, and 90 days after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 27 | 27
pg/ml
  RANKL 7 days after HCT: number analyzed (Participants) | 26 | 24
  RANKL 7 days after HCT | 58.9 (72.4) | 40.5 (36.3)
  RANKL 14 days after HCT: number analyzed (Participants) | 23 | 26
  RANKL 14 days after HCT | 45.5 (64.6) | 42.1 (44.7)
  RANKL 21 days after HCT: number analyzed (Participants) | 27 | 22
  RANKL 21 days after HCT | 49.3 (55.8) | 51.0 (48.6)
  RANKL 90 days after HCT: number analyzed (Participants) | 25 | 24
  RANKL 90 days after HCT | 56.6 (65.8) | 41.4 (27.5)
  OPG 7 days after HCT: number analyzed (Participants) | 26 | 27
  OPG 7 days after HCT | 489 (454) | 564 (315)
  OPG 14 days after HCT: number analyzed (Participants) | 25 | 26
  OPG 14 days after HCT | 617 (651) | 650 (378)
  OPG 21 days after HCT: number analyzed (Participants) | 25 | 23
  OPG 21 days after HCT | 582 (646) | 575 (290)
  OPG 90 days after HCT: number analyzed (Participants) | 24 | 25
  OPG 90 days after HCT | 499 (589) | 422 (231)

6. Secondary Outcome: Marker of Bone Resorption (Carboxy-terminal Collagen Crosslinks [CTX]
Description: CTX measured in ng/ml.
Time Frame: 7, 14, 21, 90, 180, 360 days after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 28 | 27
ng/ml
  CTX 7 days after HCT | 0.596 (0.833) | 0.455 (0.440)
  CTX 14 days after HCT: number analyzed (Participants) | 26 | 26
  CTX 14 days after HCT | 0.341 (0.165) | 0.347 (0.185)
  CTX 21 days after HCT: number analyzed (Participants) | 27 | 23
  CTX 21 days after HCT | 0.332 (0.085) | 0.441 (0.372)
  CTX 90 days after HCT: number analyzed (Participants) | 25 | 25
  CTX 90 days after HCT | 0.327 (0.117) | 0.328 (0.113)
  CTX 180 days after HCT: number analyzed (Participants) | 16 | 15
  CTX 180 days after HCT | 0.395 (0.236) | 0.318 (0.106)
  CTX 360 days after HCT: number analyzed (Participants) | 15 | 13
  CTX 360 days after HCT | 0.291 (0.119) | 0.307 (0.088)

7. Secondary Outcome: Markers of Bone Formation (Procollagen Type 1 N-terminal Propeptide [P1NP])
Description: P1NP measured in ng/ml.
Time Frame: 7, 14, 21, 90, 180, 360 days after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 28 | 27
ng/ml
  P1NP 7 days after HCT | 36.2 (14.9) | 38 (18.6)
  P1NP 14 days after HCT: number analyzed (Participants) | 26 | 26
  P1NP 14 days after HCT | 36.9 (16.8) | 35.7 (14.2)
  P1NP 21 days after HCT: number analyzed (Participants) | 27 | 23
  P1NP 21 days after HCT | 38.5 (16.4) | 37.1 (15.4)
  P1NP 90 days after HCT: number analyzed (Participants) | 25 | 25
  P1NP 90 days after HCT | 41.2 (17.9) | 39.5 (17.8)
  P1NP 180 days after HCT: number analyzed (Participants) | 16 | 15
  P1NP 180 days after HCT | 29.2 (13.7) | 27.6 (11.8)
  P1NP 360 days after HCT: number analyzed (Participants) | 15 | 13
  P1NP 360 days after HCT | 28.6 (14.5) | 29.3 (12.8)

8. Secondary Outcome: Ratio of Receptor Activator of the Nuclear Factor-κB Ligand [RANKL] and Osteoprotegerin [OPG]
Time Frame: 7 days, 14 days, 21 days, and 90 days after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 25 | 26
ratio
  RANKL/OPG 7 days after HCT: number analyzed (Participants) | 24 | 24
  RANKL/OPG 7 days after HCT | 0.154 (0.186) | 0.096 (0.103)
  RANKL/OPG 14 days after HCT: number analyzed (Participants) | 22 | 26
  RANKL/OPG 14 days after HCT | 0.10 (0.137) | 0.078 (0.085)
  RANKL/OPG 21 days after HCT: number analyzed (Participants) | 25 | 22
  RANKL/OPG 21 days after HCT | 0.121 (0.139) | 0.095 (0.086)
  RANKL/OPG 90 days after HCT: number analyzed (Participants) | 24 | 24
  RANKL/OPG 90 days after HCT | 0.205 (0.278) | 0.127 (0.109)

9. Secondary Outcome: Marker of Bone Resorption Deoxypyridinoline [DPD])
Description: DPD measured in mmol/L.
Time Frame: 7, 14, 21, 90, 180, 360 days after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 28 | 27
mmol/L
  DPD 7 days after HCT | 133 (113) | 89.7 (58.8)
  DPD 14 days after HCT: number analyzed (Participants) | 24 | 27
  DPD 14 days after HCT | 71.4 (65.7) | 70.7 (58.7)
  DPD 21 days after HCT: number analyzed (Participants) | 24 | 23
  DPD 21 days after HCT | 91.6 (78.8) | 112 (103)
  DPD 90 days after HCT: number analyzed (Participants) | 19 | 27
  DPD 90 days after HCT | 170 (130) | 146 (108)
  DPD 180 days after HCT: number analyzed (Participants) | 19 | 20
  DPD 180 days after HCT | 191 (119) | 163 (107)
  DPD 360 days after HCT: number analyzed (Participants) | 16 | 14
  DPD 360 days after HCT | 123 (87) | 145 (121)

10. Secondary Outcome: Marker of Bone Formation Osteocalcin [OCN])
Description: OCN measured in pg/ml.
Time Frame: 7, 14, 21, 90, 180, 360 days after HCT
Population: Participants unable to be evaluated due to declining health or failure of follow up.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Pamidronate Group
Number analyzed (Participants) | 26 | 27
pg/ml
  OCN 7 days after HCT | 56832 (31576) | 59071 (31740)
  OCN 14 days after HCT: number analyzed (Participants) | 25 | 26
  OCN 14 days after HCT | 57611 (37994) | 68137 (41600)
  OCN 21 days after HCT: number analyzed (Participants) | 25 | 23
  OCN 21 days after HCT | 59890 (37398) | 58983 (42097)
  OCN 90 days after HCT: number analyzed (Participants) | 24 | 25
  OCN 90 days after HCT | 48839 (33380) | 57638 (34727)
  OCN 180 days after HCT: number analyzed (Participants) | 16 | 15
  OCN 180 days after HCT | 47077 (45972) | 47459 (18955)
  OCN 360 days after HCT: number analyzed (Participants) | 15 | 16
  OCN 360 days after HCT | 85950 (126169) | 52972 (25938)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group | Pamidronate Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 9/32 | 19/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=32) | Pamidronate Group (N=31)
Heart palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Redness of the eye (Eye disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 2 (3)
Photophobia (Eye disorders) | 0 (0) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (9)
Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02074631/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT02074631/ICF_001.pdf